CLINICAL TRIAL: NCT03187483
Title: Do Adhesive Flash-free Brackets Affect Bacterial Plaque? A Randomized Controlled Clinical and Microbiological Assessment
Brief Title: Flash-free Brackets and Dental Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nurcan Buduneli, Professor, Ege University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 13-11.1/9
Record Dates: First submitted 2017-06-10; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Orthodontic Treatment
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flash-free bracket group (Active Comparator): Orthodontic treatment with flash-free bracket system
  Interventions: Procedure: orthodontic treatment
- Control (Active Comparator): Orthodontic treatment with conventional adhesive-coated brackets
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Procedure: orthodontic treatment — orthodontic treatment in maxillary crowding

SUMMARY:
This study aimed to compare flash-free bracket system with conventional adhesive-coated bracket system in patients with maxillary crowding.

DETAILED DESCRIPTION:
Aim: The aim of this split-mouth study was to compare conventional and adhesive flash-free-bracket systems in terms of plaque retention, white spot lesion formation, biomarker levels and select microbes in gingival crevicular fluid (GCF).

Materials & Methods: Thirty-seven systemically healthy patients (18 males, 19 females) with the age range of 13-18 years were involved in this split-mouth study. Clinical evaluations, quantitative light-induced fluorescence (QLF) imaging, GCF and plaque samplings were performed at baseline and at 1-, 2-, 3-months. QLF was repeated following debonding, GCF samples were analyzed by immunoassay and real-time PCR for the biomarker and bacteria content. Data were analyzed by Wilcoxon on dependent samples.

ELIGIBILITY:
Inclusion Criteria:

* being systemically healthy
* having 4-7 mm maxillary crowding with a maximum of 2 mm linear displacement of contact points and non-extraction treatment planning.

Exclusion Criteria:

-

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
development of white spot lesion (WSL) | 1 month
  WSL is the first sign of caries

SECONDARY OUTCOMES:
plaque accumulation around the brackets | 1 month
  plaque deposits cause gingival inflammation
microbial composition around the brackets | 1 month
  presence of pathogen bacteria is important

IPD SHARING:
Plan to Share IPD: No